CLINICAL TRIAL: NCT03463733
Title: International Multicenter Phase I Trial of Hydroxyurea in Combination With Dose-Intense Temozolomide in Recurrent Glioblastoma
Brief Title: Hydroxy-urea and Temozolomide in Patients With a Recurrent Malignant Brain Tumor (Glioblastoma)
Acronym: HUTMZ
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: M.E. van Linde (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor-Investigator, M.E. van Linde, MD, Principal Investigator, Amsterdam UMC, location VUmc
Organization: Amsterdam UMC, location VUmc (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro-16/11
Record Dates: First submitted 2018-03-01; First posted 2018-03-13 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Glioma; Glioblastoma
Keywords: Glioma; Recurrent glioma; Glioblastoma multiforme; Recurrent Glioblastoma multiforme; Hydroxyurea; Temozolomide
MeSH Terms: conditions — Glioma; Glioblastoma | interventions — Hydroxyurea; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Daily hydroxyurea and temozolomide (Experimental): Hydroxyurea and temozolomide will be administered every 4 weeks, with 28 consecutive days defined as a treatment cycle. Treatment will be administered on an outpatient basis. Oral hydroxyurea (dose specified by the Dose Cohort below) and oral temozolomide (50 mg/m2/day) will be administered daily in 28-day cycles for 12 cycles or until unacceptable toxicity, intolerance, progressive disease, or withdrawal of consent. Patients will be treated in dose cohorts of 3 with each cohort receiving a specific daily dose assignment of hydroxyurea.
  All patients in the study will receive temozolomide at 50 mg/m2/day ("dose-intense" schedule). The starting dose level for hydroxyurea will be 200 mg daily (QD) up to a maximum of 2000mg hydroxyurea a day.
  Interventions: Drug: Hydroxyurea; Drug: Temozolomide

INTERVENTIONS:
Drug: Hydroxyurea — 147-94-4/HYDROXYCARBAMIDE/HYDROXYCARBAMIDE/based on myeloproliferative disorders (MPD) record: SUB08076MIG
  Other Names: Hydroxycarbamide
Drug: Temozolomide — 85622-93-1 /TEMOZOLOMIDE/TEMOZOLOMIDE/based on myeloproliferative disorders (MPD) record: SUB10889MIG
  Other Names: Temodar

SUMMARY:
Background

Currently, no standard treatment exists for patients with recurrent glioblastoma multiforme (rGBM) and used 2nd line treatments have low (up to max. 20%) response rates and very modest response duration (months). The median overall survival for GBM patients is 12-14 months from the time of diagnosis; therefore the development of new therapeutic options is imperative. HU has been used to treat hematological diseases and solid tumors (such as melanoma, ovarian, squamous cell carcinoma, head and neck carcinoma and brain tumors) in combination with other anti-cancer agents, but never with TMZ. If found safe, HU+TMZ, is easily translated to the clinic.

Purpose: Phase I trial to identify the maximum tolerated dose (MTD) for the combination of dose intense temozolomide (TMZ) and hydroxy-urea (HU) in (maximal) thirty patients with recurrent glioblastoma (rGBM).

Plan of investigation:

Month 0-24 (1st and 2nd year): Inclusion and follow-up of a maximum of 30 patients with rGBM

Month 25-31 (3rd year): Follow-up of patients included in the trial, data analysis (determining MTD and explorative analysis) and manuscript preparation.

Possible results:

1. Obtaining MTD and safety profile of daily HU+TMZ in patients with rGBM;
2. Preliminary data on the estimation of the median progression-free (PFS) and overall survival (OS), radiographic response proportion in patients with measurable disease, and exploratory correlation of treatment outcomes (PFS and OS) with o6-methylguanine-DNA-methyltransferase (MGMT) promoter methylation status in archival tumor specimens and further elucidation of underlying mechanism of re-sensitization of TMZ by HU. Exploratory analysis of biomarkers profile of platelets in patients treated with HU+TMZ.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have histologically or cytologically confirmed glioblastoma multiforme
2. Patients may have had any number of prior therapies for glioblastoma. Patients must be at least 28 days from any investigational agent, 28 days from prior cytotoxic therapy (except 23 days from prior temozolomide, 14 days from vincristine, 42 days from nitrosoureas, 21 days from procarbazine administration), and 7 days for patients who received metronomic chemotherapy or non-cytotoxic agents, e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid, etc.
3. Age ≥18 years. Because no dosing or adverse event data are currently available on the use of hydroxyurea in combination with temozolomide in participants <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
4. Karnofsky Performance Status (KPS) ≥60%
5. Participants must have normal organ and marrow function as defined below:

   * leukocytes ≥3,000/microliter (mcL)
   * absolute neutrophil count ≥1,500/mcL
   * platelets ≥100,000/mcL
   * total bilirubin within normal institutional limits
   * Aspartate transaminase (AST; SGOT)/alanine transaminase (ALT; SGPT) ≤2.5 × institutional upper limit of normal
   * creatinine below upper limit of normal institutional limits OR
   * creatinine clearance ≥60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
6. Progressive disease on contrast-enhanced brain CT or MRI as defined by Response Assessment in Neuro-Oncology (RANO) Criteria [22], or have documented recurrent glioblastoma on diagnostic biopsy. Patients who have been previously treated with bevacizumab therapy that have T2-weighted or FLAIR MRI sequences considered to be progressive disease by the study investigator but have no contrast-enhancing areas of recurrent disease are eligible.
7. Interval of at least 2 weeks from any prior neurosurgical resection (1 week for intracranial biopsy) to start of study drug; and patient must have adequate wound healing.
8. Interval of at least 12 weeks from prior radiotherapy unless there is either: a) histopathologic confirmation of recurrent tumor, or b) new enhancement on MRI outside of the radiation treatment (RT) field.
9. Because cytotoxic agents such as temozolomide and hydroxyurea are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of temozolomide and hydroxyurea administration.
10. Patients must have archival tumor tissue available for molecular analysis and must be willing to consent for this tissue to be analyzed as part of this study. However, if no archival tumor tissue is available, the patient will not be excluded from the study.
11. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Participants who are receiving any other investigational agents or devices in investigation for glioblastoma.
2. Patients must not have been previously treated with an anti-vascular endothelial growth factor (VEGF) inhibitor.
3. History of allergic reactions attributed to compounds of similar chemical composition to temozolomide and/or hydroxyurea.
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
5. Pregnant women are excluded from this study because hydroxyurea and temozolomide have known teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with hydroxyurea and temozolomide, breastfeeding should be discontinued if the mother is treated with hydroxyurea and temozolomide.
6. HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with hydroxyurea. In addition, these participants are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
7. Patients with a history of a different malignancy are ineligible except for the following circumstances: if they have been disease-free for at least 3 years and are deemed by the investigator to be at low risk for recurrence of that malignancy; patients with treated cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin. Patients will not be eligible if they have evidence of other malignancy requiring therapy other than surgery within the last 3 years.
8. Major surgery (not including minor diagnostic procedures such as lymph node biopsy) within 2 weeks of start of study drug; or not fully recovered from any side effects of previous procedures.
9. Presence of extra-cranial metastatic disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2018-03-02 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Maximal tolerated dose (MTD) hydroxyurea in combination with dose intense temozolomide | 12 months
  MTD

CONTACTS AND LOCATIONS:
Overall Officials: ME van Linde, MD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
In anonymized form